CLINICAL TRIAL: NCT07132775
Title: Evaluation of the Safety and Efficacy of a Full-Body Electrostimulation Garment for Individuals With Neurological and Neuromuscular Conditions That Cause Spasticity, Hyperreflexia, and Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Collaborators: Otto Bock Healthcare Products GmbH (Industry)
Responsible Party: Principal Investigator, Arun Jayaraman, PT, PhD, Director - Max Nader Center for Rehabilitation Technologies and Outcomes Research, Shirley Ryan AbilityLab
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: STU00221544
Record Dates: First submitted 2025-07-23; First posted 2025-08-20 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Multiple Sclerosis; Fibromyalgia; Neurologic Disorder; Neuromuscular Disorders
MeSH Terms: conditions — Multiple Sclerosis; Fibromyalgia; Nervous System Diseases; Neuromuscular Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Intervention (Experimental): Participants will wear the full-body electrostimulation garment for 60 minutes at a time, every other day, with the stimulation parameters actively running.
  Interventions: Device: Active full-body stimulation
- Sham (Sham Comparator): Participants will wear the full-body electrostimulation garment for 60 minutes at a time, every other day, with the stimulation parameters not actively running.
  Interventions: Other: Sham full-body stimulation

INTERVENTIONS:
Device: Active full-body stimulation — Participants will receive active stimulation through a full-body suit with embedded electrodes that deliver a low-grade electrical stimulation to muscle groups.
  Arms: Intervention
Other: Sham full-body stimulation — Participants will receive sham stimulation through a full-body suit with embedded electrodes that deliver a low-grade electrical stimulation to muscle groups.
  Arms: Sham

SUMMARY:
The purpose of this study is to to explore the safety and efficacy of the EXOPULSE Mollii suit, a full-body electrostimulation suit, for individuals with neurological or neuromuscular conditions that cause spasticity, hyperreflexia, and/or pain.

DETAILED DESCRIPTION:
Optimization Aim: Identify a systematic, methodological approach to device fitting, inclinic and at-home protocols using the Mollii suit, and optimization of collecting outcome measures at assessment visits. For example, up to 15 participants will complete a portion or all of the procedures listed in the "Procedures Involved" section of this protocol to determine an optimal approach.

Aim 1: Assess the safety of the Mollii suit during an in-clinic or at-home 12-week period consisting of daily sessions of a 60-minute duration in individuals with pain and/or spasticity from neurological and neuromuscular conditions that cause spasticity, hyperreflexia, and pain.

Aim 2: Evaluate the use of full-body active electrostimulation as compared to full-body sham electrostimulation as an intervention in-clinic or at-home for individuals experiencing pain and/or spasticity due to neurological and neuromuscular conditions that cause spasticity, hyperreflexia, and pain.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 75 years old
2. Medical clearance from physician
3. Individuals who experience spasticity, pain, or hyperreflexia due to neurological or neuromuscular conditions or individuals with a diagnosis of Multiple Sclerosis or Fibromyalgia
4. For participants with a diagnosis of Multiple Sclerosis:

   1. having a definite diagnosis for at least one month
   2. Ability to walk independently or with the need of support (expanded disability status scale score (EDSS) < 7).
   3. Absence of relapses in the last three months
   4. Demonstrating spasticity with a score of at least 1+ on the Modified Ashworth Scale (MAS)
   5. Berg Balance Scale (BBS) score of < 46 (associated in the literature with a risk of fall)
5. For participants with a diagnosis of Fibromyalgia:

   a. having a definite diagnosis for at least three months
6. Able to follow instructions and inform study staff of pain and/or discomfort
7. Able to ambulate 10m without body weight support with or without assistive devices and/or caregiver assistance

Exclusion Criteria:

1. Implanted medical devices or equipment which can be disrupted by magnets (ex. Shunts)
2. Swollen, infected, or inflamed areas or skin eruptions (e.g., phlebitis, thrombophlebitis, varicose veins, etc.) in areas where the suit will be used
3. No established somatic or neuropsychiatric diagnosis prior to enrollment in the study
4. Pregnant and/or nursing

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-07-23 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Berg Balance Scale | Baseline 1 (prior to Arm 1)- initial visit, Endpoint 1 (after 2 weeks of Arm 1)- at approx 2 weeks, Baseline 2 (after 2 week washout and before Arm 2)- at approx 4 weeks, Endpoint 2 (after 2 weeks of Arm 2)- at approx 6 weeks
  The Berg Balance Scale is a 14-item objective measure that assesses static balance and falls risk. The functional abilities that are assessed include sitting and standing balance, transfers, altered bases of support, reaching, turning, and closing eyes.Scores range from 0 - 56, with higher scores indicating improved balance.

SECONDARY OUTCOMES:
Manual Muscle Test | Baseline 1 (prior to Arm 1)- initial visit, Endpoint 1 (after 2 weeks of Arm 1)- at approx 2 weeks, Baseline 2 (after 2 week washout and before Arm 2)- at approx 4 weeks, Endpoint 2 (after 2 weeks of Arm 2)- at approx 6 weeks
  A procedure to evaluate the strength of individual muscles relative to gravity and manual resistance. Scores can range from 0 (no contraction) to 5 (full contraction against max resistance)
Modified Ashworth Scale | Baseline 1 (prior to Arm 1)- initial visit, Endpoint 1 (after 2 weeks of Arm 1)- at approx 2 weeks, Baseline 2 (after 2 week washout and before Arm 2)- at approx 4 weeks, Endpoint 2 (after 2 weeks of Arm 2)- at approx 6 weeks
  The Modified Ashworth Scale is used to grade the amount of hypertonicity / spasticity in individuals. Tone is scored by passively moving the individual's limb and assessing the amount of resistance to movement felt by the examiner. Scores can range from 0 (no spasticity) to 4 (affected part rigid.)
10 Meter Walk Test | Baseline 1 (prior to Arm 1)- initial visit, Endpoint 1 (after 2 weeks of Arm 1)- at approx 2 weeks, Baseline 2 (after 2 week washout and before Arm 2)- at approx 4 weeks, Endpoint 2 (after 2 weeks of Arm 2)- at approx 6 weeks
  Participants are timed as they walk 10 meters at both their self-selected speed, and their fastest but safest speeds.
6 Minute Walk Test | Baseline 1 (prior to Arm 1)- initial visit, Endpoint 1 (after 2 weeks of Arm 1)- at approx 2 weeks, Baseline 2 (after 2 week washout and before Arm 2)- at approx 4 weeks, Endpoint 2 (after 2 weeks of Arm 2)- at approx 6 weeks
  A test to measure the distance that a participant can walk over a period of 6 minutes.
Timed Up and Go | Baseline 1 (prior to Arm 1)- initial visit, Endpoint 1 (after 2 weeks of Arm 1)- at approx 2 weeks, Baseline 2 (after 2 week washout and before Arm 2)- at approx 4 weeks, Endpoint 2 (after 2 weeks of Arm 2)- at approx 6 weeks
  The Timed Up and Go measures the time it takes for a person to stand up from a chair, walk a distance of 3 meters, turn, walk back to the chair, and sit down.
Twelve-Item Multiple Sclerosis Walking Scale | Baseline 1 (prior to Arm 1)- initial visit, Endpoint 1 (after 2 weeks of Arm 1)- at approx 2 weeks, Baseline 2 (after 2 week washout and before Arm 2)- at approx 4 weeks, Endpoint 2 (after 2 weeks of Arm 2)- at approx 6 weeks
  A self-report questionnaire that measures the impact of multiple sclerosis on a person's walking ability. Scores range from 12 - 60, with higher scores indicating a greater impact on walking ability.
Falls Efficacy Scale | Baseline 1 (prior to Arm 1)- initial visit, Endpoint 1 (after 2 weeks of Arm 1)- at approx 2 weeks, Baseline 2 (after 2 week washout and before Arm 2)- at approx 4 weeks, Endpoint 2 (after 2 weeks of Arm 2)- at approx 6 weeks
  A questionnaire that measures a participant's fear of falling for items related to activities of daily living. Scores range from 10 - 100, with higher scores indicating an increased fear of falling.
Multiple Sclerosis International Quality of Life Questionnaire | Baseline 1 (prior to Arm 1)- initial visit, Endpoint 1 (after 2 weeks of Arm 1)- at approx 2 weeks, Baseline 2 (after 2 week washout and before Arm 2)- at approx 4 weeks, Endpoint 2 (after 2 weeks of Arm 2)- at approx 6 weeks
  A multi-dimensional questionnaire about a patient's quality of life for those who have multiple sclerosis.
Clinical Global Impressions Scale | Baseline 1 (prior to Arm 1)- initial visit, Endpoint 1 (after 2 weeks of Arm 1)- at approx 2 weeks, Baseline 2 (after 2 week washout and before Arm 2)- at approx 4 weeks, Endpoint 2 (after 2 weeks of Arm 2)- at approx 6 weeks
  A assessment of the clinician's view of a participant's global functioning prior to, and after initiating a study intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Shirley Ryan AbilityLab, Chicago, Illinois, United States